CLINICAL TRIAL: NCT01595893
Title: Vitamin D3 Supplementation in Polymorphic Light Eruption: Randomized Double-blinded Placebo-controlled Trial
Brief Title: Vitamin D Supplementation in Polymorphic Light Eruption
Acronym: VitD-PLE_2012
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Difficulties in recruiting the planned number of patients
Sponsor: Medical University of Graz (Other)
Collaborators: Austrian Science Fund (FWF) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Graz 24-220 ex 11/12
Record Dates: First submitted 2012-04-26; First posted 2012-05-10 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-06

CONDITIONS: Polymorphic Light Eruption
Keywords: Polymorphic light eruption; Vitamin D3; Photo provocation; Immune function
MeSH Terms: interventions — Cholecalciferol; Plant Oils

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D3 (Experimental)
  Interventions: Drug: Oral Vitamin D 3
- Placebo (Placebo Comparator)
  Interventions: Drug: Miglyol 812 N

INTERVENTIONS:
Drug: Oral Vitamin D 3 — 40,000 IE vitamin D3 per 70 kg body weight, given twice (2 weeks apart)
  Other Names: Oleovit D3, Fresenius Kabi, Austria
  Arms: Vitamin D3
Drug: Miglyol 812 N — Neutral oil of esters extracted from coconut and palm kernel
  Other Names: Vegetable oil
  Arms: Placebo

SUMMARY:
Polymorphic light eruption (PLE) is a common photodermatosis with a high prevalence of approximately 11 to 21% in the population. Similar to lupus erythematosus (LE), an UV-inducible systemic autoimmune disease, PLE has a female preponderance with a mean onset in the second to third decade of life. PLE lesions are very itchy and typically appear on sun-exposed body sites in spring or early summer. The quality of life in patients with PLE is often severely disturbed, as evidenced by high levels of anxiety and depression. For prophylaxis besides conventional sunscreens, photo(chemo)therapy is effective in many cases, when administered over several weeks for hardening in early spring before the first natural sun exposure takes place. However, because prolonged treatment with UVB and/or photochemotherapy is potentially carcinogenic, the search for pathogenic mechanisms and new treatment options in PLE is ongoing. The exact pathogenesis of PLE is currently unknown but findings suggest an autoimmune-type background with resistance to UV-induced immune suppression and simultaneous immune reactions against skin photo-neoantigens. The investigators have recently found that PLE patients had significantly reduced 1,25-(OH)2-vitamin D3 serum levels (13-14ng/ml) compared to the normal population (>30ng/ml). In addition, the investigators were able to demonstrate in an intra-individual half-body trial that topical administration of an immunostimulatory 1,25-(OH)2-vitamin-D3 analogue calcipotriol reduced PLE symptoms in an experimental study. In the proposed randomized double-blinded placebo-controlled trial the investigators attempt to study the effect of oral vitamin D3 supplementation (2 x 40.000 IE, given orally two weeks apart) on PLE symptoms.

DETAILED DESCRIPTION:
PLE patients will be subjected to experimental photo provocation with solar simulated UV radiation over several days before and after vitamin D3 supplementation. Disease symptoms will be quantified with a newly established and validated PLE test score, (AA + SI + 0.4P [range, 0-12], where AA is affected area score [range, 0-4], SI is skin infiltration score [range, 0-4], and P is pruritus score on a visual analogue scale [range, 0-10]). Optional biopsies will be taken to investigate the effect of oral vitamin D3 on UV-induced skin test sites, including cellular skin infiltration and expression and release of cytokines in situ as endpoints. We will also study the effect of oral vitamin D3 on abnormalities i) of levels and function of regulatory T cells, ii) chemotaxis of leucocytes, and iii) proinflammatory cytokines, i.e. alterations that have been previously linked to PLE pathogenesis. This will be done by i) FACS and co-culture T cell proliferation assays, ii) response of peripheral neutrophil leucocytes to the chemoattractants leukotriene B4 (LTB4) and formyl-methionyl-leucyl-phenylalanine, and iii) ELISA and immunobead assay of patient serum.

To back-up the results obtained with the PLE test score upon experimental photo provocation the study participants will receive a questionnaire on PLE symptoms and quality of life, adapted from scores as previously described. This questionnaire will allow monitoring PLE symptoms and quality of life in the patients during the summer season following the oral vitamin D3 supplementation in spring.

The results of the project will enlighten the mechanism of PLE and may establish the base of a novel prevention strategy via the vitamin D3 pathway.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of PLE by typical patient history, typical histology of skin lesions and/or positive photo provocation results

Exclusion Criteria:

* Allergy or intolerance to Oleovit D3 or Coconut/palm kernel
* Presence or history of malignant skin tumors
* Dysplastic melanocytic nevus syndrome
* Photosensitive diseases such as porphyria, chronic actinic dermatitis, xeroderma pigmentosum, and basal cell nevus syndrome; autoimmune disorders such as lupus erythematosus or dermatomyositis
* Sarcoid
* Renal dysfunction
* Psychiatric disorder
* Pregnancy or breastfeeding
* Topical treatment with vitamin D derivates within 3 months
* Oral treatment with vitamin D within 6 months
* Antinuclear antibodies such as anti-ds-DNA or anti- Ro/La
* 25-hydroxy vitamin D serum levels > 30ng/ml at screening visit
* Serum hypercalcemia > 2,65 nmol/L
* Treatment with thiazides or glycosides
* Systemic treatment with steroids and/or other immunosuppressive drugs within 4 weeks
* UV exposure in test fields within 8 weeks before the start of the study
* General poor health status

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
PLE test score (from 0-12) of experimental photo provocation | At day 2, 3, 4, 5, and 8 (change from baseline)
  See study description.

SECONDARY OUTCOMES:
Cytokine levels in serum | At day 22 and 36; and at month 4-8
Chemotaxis of neutrophils | At day 22 and 36; and at month 4-8 (compared to baseline)
Level of regulatory T cells | At day 22 and 36; and at month 4-8 (compared to baseline)
Quantification of skin alterations, including cellular infiltration and cytokine profile | Day 5 and 40
Dermatological quality of life (DLQI) | At month 4-8
HADS (hospital anxiety and depression scale) | At month 4-8
Function of regulatory T cells | 22 and 36; and at month 4-8 (compared to baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Wolf, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Department of Dermatology, Graz, Austria

REFERENCES:
- [Derived] Schweintzger NA, Gruber-Wackernagel A, Shirsath N, Quehenberger F, Obermayer-Pietsch B, Wolf P. Influence of the season on vitamin D levels and regulatory T cells in patients with polymorphic light eruption. Photochem Photobiol Sci. 2016 Mar;15(3):440-6. doi: 10.1039/c5pp00398a. Epub 2016 Feb 25. PMID 26911519